CLINICAL TRIAL: NCT06831422
Title: Application of a Novel Antimicrobial Wash Versus Hydrogen Peroxide Versus Povidone-iodine to the Dermis and Incidence of Cutibacterium Acnes During Shoulder Arthroplasty: A Randomized Controlled Trial
Brief Title: Post-incision Antimicrobial Wash vs C. Acnes in Shoulder Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Next Science TM (Industry)
Responsible Party: Principal Investigator, Jared Mahylis, Orthopaedic Surgeon, Prinicipal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17996
Record Dates: First submitted 2025-02-12; First posted 2025-02-18 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Shoulder Arthroplasty; Positive C. Acnes Culture
Keywords: Shoulder Arthroplasty; Antimicrobial; Post-incision wash; C. Acnes
MeSH Terms: interventions — Arthroplasty, Replacement, Shoulder

STUDY DESIGN:
Intervention Model Description: All groups will receive standard presurgical preparation with standard surgical skin preparation. This begins with each subject receiving two chlorhexidine scrub brushes with which they will be instructed to scrub themselves the night before and morning of their surgery. Once in the operating room, all subjects will have their surgical site treated with Chlorhexidine Gluconate 4% soap, once with 3% hydrogen peroxide, and then twice with standard operative skin preparation agent, Chloraprep (2% chlorhexidine gluconate (CHG) and 70% v/v isopropyl alcohol). No preoperative acetic acid, betadine, or benzoyl peroxide will be applied to the surgical shoulder. The intervention will only take place after the initial incision has been made. Subjects will be randomly assigned in a 1:1:1:1 fashion to groups that will either receive one of the wash solutions (Xperience, Povidone, or Hydrogen peroxide) or a control group that will receive no post-incision wash.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Xperience Antimicrobial Wash (Experimental): Xperience Antimicrobial Wash is composed of 32.5 g/L citric acid, 31.3 g/L sodium citrate, and 1.00 g/L sodium lauryl sulfate in sterile water. It is to be applied along the entire dermis using a soaked surgical sponge following initial incision.
  Interventions: Device: Xperience Antimicrobial Wash; Diagnostic Test: Bacterial Cultures; Procedure: Shoulder Arthroplasty
- 3% hydrogen peroxide (Experimental): To be applied along the entire dermis using a soaked surgical sponge following initial incision.
  Interventions: Device: Hydrogen Peroxide; Diagnostic Test: Bacterial Cultures; Procedure: Shoulder Arthroplasty
- 10% povidone-iodine (Experimental): To be applied along the entire dermis using a soaked surgical sponge following initial incision.
- Control (Active Comparator): No treatment of the dermal layer will be performed prior to a collection of the bacterial cultures
  Interventions: Diagnostic Test: Bacterial Cultures; Procedure: Shoulder Arthroplasty

INTERVENTIONS:
Device: Povidone-Iodine — Following electrocautery opening of the dermal layer, patients in the povidine-iodine group (Group B) will receive application of 10% sterile povidone-iodine along the entire dermis using a soaked surgical sponge. Approximately 120 seconds after application of betadine, a culture of the dermis will then be taken by dragging the culture swab along the length of the exposed dermis (dermis culture).
Device: Hydrogen Peroxide — Following electrocautery opening of the dermal layer, patients in the hydrogen peroxide group (Group A) will receive application of 3% sterile-filtered hydrogen peroxide along the entire dermis using a soaked surgical sponge. Approximately 120 seconds after application of hydrogen peroxide a culture of the dermis will then be taken by dragging the culture swab along the length of the exposed dermis (dermis culture).
  Arms: 3% hydrogen peroxide
Device: Xperience Antimicrobial Wash — Following electrocautery opening of the dermal layer, patients in the patients in the Xperience group (Group C) will receive application of the Xperience antimicrobial wash (NextScience, Jacksonville, FL) (32.5 g/L citric acid, 31.3 g/L sodium citrate, and 1.00 g/L sodium lauryl sulfate in sterile water) along the entire dermis using a soaked surgical sponge. Approximately 120 seconds after application of Xperience, a culture of the dermis will then be taken by dragging the culture swab along the length of the exposed dermis (dermis culture).
  Arms: Xperience Antimicrobial Wash
Diagnostic Test: Bacterial Cultures — Four C. Acnes cultures will be obtained for every patient. Once the skin has dried, a culture swab will be applied along the planned incision for all patients (skin culture). Approximately 120 seconds after application of Xperience, hydrogen peroxide or betadine, or after initial incision in the case of the control group, a culture of the dermis will then taken by dragging the culture swab along the length of the exposed dermis (dermis culture). Once the glenohumeral joint is exposed, the surgeon will apply new surgical gloves, and a culture swab will be placed into the joint and along the humeral head (glenohumeral joint culture). An additional culture will then be taken from the air in the operative suite (air culture)
  Arms: 3% hydrogen peroxide; Control; Xperience Antimicrobial Wash
Procedure: Shoulder Arthroplasty — All patients will undergo hemiarthroplasty, anatomic total shoulder arthroplasty, or reverse total shoulder arthroplasty in accordance with the appropriate indications and enrollment in this study.
  Arms: 3% hydrogen peroxide; Control; Xperience Antimicrobial Wash

SUMMARY:
The purpose of this randomized controlled trial is to determine the effect of post-incision wash using various novel antimicrobial solutions on the rate of positive C. Acnes cultures collected from adults undergoing primary shoulder replacement surgery. Subjects will be randomly assigned in a 1:1:1:1 fashion to groups that will receive one of the following treatments:

* Post-incision application of Xperience Antimicrobial wash (NextScience, Jacksonville, FL)
* Post-incision application of 3% hydrogen peroxide
* Post-incision application of 10% povidone-iodine (betadine)
* No post-incision treatment (control)

The investigators hypothesize that the subjects treated with the antimicrobial solutions after initial incision will have lower rates of positive C. Acnes cultures. The investigators also hypothesize that post-incision application of Xperience Antimicrobial wash and Betadine will have an equal reduction in the incidence of C. acnes as Hydrogen Peroxide.

DETAILED DESCRIPTION:
Cultures will be collected from the following sites:

* The surgical site prior to the initial incision
* The incision site after the initial incision
* The shoulder joint
* The room air

Cultures will be monitored daily for the presence of C. Acnes up to 18 days post-surgery. At postoperative clinic visits, patients in all groups will undergo a clinical evaluation by their surgeon, which includes assessment of wound healing and any complications at 2 weeks, 6 weeks, 3 months, 6 months, and 1 year following surgery. A password-secured database and data points will be pulled from electronic medical records. Data will be analyzed and will be utilized to come to the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Indicated and scheduled for primary shoulder arthroplasty.
* Chronic severe glenohumeral osteoarthritis, avascular necrosis, post traumatic osteoarthritis, rotator cuff arthropathy,
* Ability to read and understand English
* Age ≥18 years
* Patient failed ≥6 weeks of conservative treatment, which included non-steroidal anti-inflammatory drugs (NSAIDS)

Exclusion Criteria:

* Patient with history of prior native shoulder septic arthritis or infection
* Prior surgery of affected shoulder
* Proximal Humerus Fracture
* Active infection
* Cancer
* Autoimmune and rheumatologic disorders, including rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus
* History of allergic reaction to citric acid-derived products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of C. Acnes | up to 18 days
  C. Acnes cultures will be sampled from surgical site prior to the initial incision (skin culture), from the incision site after the initial incision (dermal culture), from the glenohumeral joint (glenohumeral joint culture), and from the room air (air culture). Each culture will be monitored for up to 18 days for growth of C. Acnes.

SECONDARY OUTCOMES:
Number and Types of Complications | up to 1 year postop.
  Patients will be closely monitored for intraoperative and postoperative complications and any sign of adverse reactions to these solutions.
Number of Subjects that Require Postoperative Reoperations | up to 1 year postop
  Whether or not patients require another operation will be documented. The number of patients requiring postoperative reoperation will be compared between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers